CLINICAL TRIAL: NCT04486365
Title: Bifocal Versus Trifocal External Bone Transport by Ilizarov Ring External Fixator as a Treatment Method for Posttraumatic Bone Defects More Than 5cm in Lower Extremities in Adults
Brief Title: Bifocal vs Trifocal External Bone Transport by Ilizarov Ring External Fixator in Lower Limbs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Mohsen Mohammed Ahmed, Resident physician in orthopedic surgery department., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ilizarov ring external fixator
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Bone Loss
Keywords: bone transport / ilizarov ring external fixator
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bifocal bone transport (Active Comparator): The bifocal approach is a single osteotomy to create one transported bone segment between the osteotomy and the defect.
  Interventions: Procedure: Bifocal bone transport.
- Trifocal bone transport (Active Comparator): The trifocal approach is two osteotomies creating two separate transported bone segments between osteotomy and defect.
  Interventions: Procedure: Trifocal bone transport

INTERVENTIONS:
Procedure: Bifocal bone transport. — The bifocal approach is a single osteotomy to create one transported bone segment between the osteotomy and the defect.
  Arms: Bifocal bone transport
Procedure: Trifocal bone transport — The trifocal approach is two osteotomies creating two separate transported bone segments.
  Arms: Trifocal bone transport

SUMMARY:
To compare between bifocal and trifocal external bone transport by ilizarov ring external fixator as a treatment method for posttraumatic bone defects more than 5cm in lower extremities regarding:

* External fixation index .
* The need of any further surgical procedures as debridement at docking site , the need of cancellous bone graft or the use of internal fixation.
* Functional outcome, complication rate as well as limb length discrepancy.

DETAILED DESCRIPTION:
Distraction osteogenesis is formation of new bone(regenerate bone) when bone segments undergo gradual, controlled separation.

There are three treatment approaches by ilizarov ring external fixator according to number of bone osteotomies. First one is the monofocal approach with closure of defect without any osteotomies. Second one is the bifocal approach with a single osteotomy to create one transported bone segment between the osteotomy and the defect. Third one is the trifocal approach with two osteotomies creating two separate transported bone segments.

Hypothetically, trifocal approach has shorter treatment time than bifocal one as it is a double level bone transport so closes the defect faster. However, there are other considerations as complications that may occur and the need of further surgical procedures and this is what will be discussed in this research.

ELIGIBILITY:
Inclusion Criteria:

* 1)Age from 18-60ys . 2)Posttraumatic bone defects more than 5 cm. 3)Lower extremity bone defects.

Exclusion Criteria:

* 1)Young pts <18 or old pts>60. 2)Post infectious or post-resection of a tumor bone defects. 3)Upper extremity bone defects.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
External fixation index | 12 to 15 months
  the number of days the external fixator is attached to the bone per centimeter of length gained.

REFERENCES:
- [Background] Hansen M, Mehler D, Voltmer W, Rommens PM. [The extraarticular proximal tibial fractures]. Unfallchirurg. 2002 Oct;105(10):858-72. doi: 10.1007/s00113-002-0529-x. German. PMID 12376892
- [Background] Court-Brown CM, Caesar B. Epidemiology of adult fractures: A review. Injury. 2006 Aug;37(8):691-7. doi: 10.1016/j.injury.2006.04.130. Epub 2006 Jun 30. PMID 16814787
- [Background] Gaebler C, Berger U, Schandelmaier P, Greitbauer M, Schauwecker HH, Applegate B, Zych G, Vecsei V. Rates and odds ratios for complications in closed and open tibial fractures treated with unreamed, small diameter tibial nails: a multicenter analysis of 467 cases. J Orthop Trauma. 2001 Aug;15(6):415-23. doi: 10.1097/00005131-200108000-00006. PMID 11514768
- [Background] Giannoudis PV, Papakostidis C, Roberts C. A review of the management of open fractures of the tibia and femur. J Bone Joint Surg Br. 2006 Mar;88(3):281-9. doi: 10.1302/0301-620X.88B3.16465. No abstract available. PMID 16497997